CLINICAL TRIAL: NCT06633432
Title: Postoperative Sleep Quality and Pain of Patients After Video-Assisted Thoracoscopic Surgery
Acronym: PSQ
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, LIna Huang, Chief Physician of Anesthesiology Department, Shanghai General Hospital, Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Yuan Lun Shen 【2024】No.164
Record Dates: First submitted 2024-09-28; First posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Sleep Disorder
MeSH Terms: conditions — Sleep Wake Disorders | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Using SPSS 25.0 software, random numbers from 001 to 316 were generated through a computer and randomly assigned in a 1:1 ratio to either the acupuncture group or the sham acupuncture group. The group information is sealed in opaque envelopes numbered randomly. Qualified subjects will be randomly assigned numbers in descending order of enrollment, without skipping numbers. Before implementing acupuncture and moxibustion, the acupuncture and moxibustion shall open the envelope allocated with the corresponding random number of the subject and conduct acupuncture and moxibustion according to the grouping information in the envelope. However, there was no communication between the acupuncture and moxibustion and other researchers and study patients about this study. Patients, attending anesthesiologists, surgeons, and data collectors (doctors responsible for evaluating sleep variables in the sleep laboratory) are all unaware of group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture group (Experimental): The acupuncture group administered medication three times at each acupoint: (1) the night before surgery, (2) the night of surgery, and (3) the first night after surgery. Acupuncture and moxibustion stimulation was applied to four pairs of acupoints: bilateral Shenmen (HT7), Neiguan (PC6), Zusanli (ST36) and Zhaohai (KI6), and the penetration depth was 10-20mm. Select the specific depth based on the subject's body type (tall, short, fat, thin). After the puncture, the acupuncture and moxibustion lifted and twisted the needle handle, and then retained the needle for 20 minutes.
  Interventions: Other: Acupuncture
- Sham-acupuncture group (Sham Comparator): The sham acupuncture group received non skin breaking comfort needles at corresponding points for acupuncture and moxibustion the night before the operation, the night of the operation and the first night after the operation, and kept the needles for 20 minutes. Non transdermal comfort needles can cause patients to experience a "needle like sensation" similar to piercing the skin, but in reality, they do not break the skin.
  Interventions: Other: Sham-acupuncture stimulation

INTERVENTIONS:
Other: Acupuncture — Administer medication at each acupoint a total of three times: (1) the night before surgery, (2) the night of surgery, and (3) the first night after surgery. In the acupuncture group, the acupuncture and moxibustion successively acupunctured four points with a depth of 10-20mm. Select the specific depth based on the subject's body type (tall, short, fat, thin). After the puncture, the acupuncture and moxibustion lifted and twisted the needle handle, and then retained the needle for 20 minutes.
  Arms: Acupuncture group
Other: Sham-acupuncture stimulation — The sham acupuncture group received non skin breaking comfort needles at the corresponding points for acupuncture and moxibustion and retained the needles for 20 minutes. Non transdermal comfort needles can cause patients to experience a needle like sensation similar to piercing the skin, but in reality, they do not break the skin.
  Other Names: sham acupuncture
  Arms: Sham-acupuncture group

SUMMARY:
The goal of this clinical trial is to to explore the effect of perioperative transcutaneous acupoint acupuncture and moxibustion stimulation on sleep quality and postoperative chronic pain in patients undergoing thoracoscopic assisted radical resection of lung cancer, and explore its potential mechanism. This clinical trial focus on the following questions:

Whether perioperative transcutaneous acupoint acupuncture and moxibustion stimulation reduce the incidence of Postoperative Sleep Disorder and postoperative acute and chronic pain ? What medical problems do participants have when taking acupuncture? Researchers will compare acupuncture to sham acupuncture (Non transdermal comfort needles can cause patients to experience a needle like sensation; similar to when the needle is inserted into the skin, but in reality, it does not break the skin) to see if acupuncture works to reduce the incidence of Postoperative Sleep Disorder and postoperative acute and chronic pain.

Participants will:

Take acupuncture or a sham acupuncture every day for 3 days(the night before surgery, the night of surgery and the first night after surgery).

On the day before surgery, the first day after surgery, the second day after surgery, and the day before discharge, the sleep status should be continuously monitored using a sleep monitoring screening device (ZG-S01D) The incidence of pain is determined by whether there is pain (including all discomfort) during patient follow-up.

DETAILED DESCRIPTION:
This experiment is divided into two groups: the experimental group and the control group. If you participate in the experiment, you will be randomly assigned to two groups, with a 50% probability of entering the experimental group and a 50% probability of entering the control group.

Research steps Anesthesia process i. Preoperative preparation Complete the scoring form, continuous dynamic blood pressure monitoring, and continuous electrocardiogram monitoring 24 hours before surgery. All patients were fasted and deprived of water for 8 hours before surgery. The upper limb venous access was opened in the pre anesthesia room. Bupivacaine liposomes were used to block the intercostal nerves in 4 intercostal spaces above and below the incision, and invasive anesthesia was performed around the surgical incision and drainage tube placement. Supplement sodium lactate Ringer solution according to the preoperative loss amount. Confirm the informed consent status again.

After entering the room, routine electrocardiographic monitoring (ECG), non-invasive arterial blood pressure (NIBP), oxygen saturation (SpO2), and mask oxygen inhalation were performed.

ii. Anesthesia induction and maintenance Anesthesia induction: Inject sufentanil 0.4ug/kg and propofol 1.5-2mg/ml intravenously in sequence. After the patient's consciousness disappears, inject rocuronium 0.6mg/kg intravenously, insert a double lumen bronchial tube (F35-37), and locate with a fiberoptic bronchoscope.

Anesthesia maintenance: maintained by inhalation of sevoflurane, intraoperative detection of end tidal sevoflurane MAC value, maintained at 1.0-1.2MAC; Administer sufentanil and rocuronium bromide intravenously as needed during surgery.

Anesthesia recovery: The patient is transferred to the post anesthesia care unit (PACU) after conscious extubation, and then transferred to the ward to ensure complete consciousness. The Aldrete score is ≥ 9.

Treatment and follow-up process i. The acupuncture group administered medication three times at each acupoint: (1) the night before surgery, (2) the night of surgery, and (3) the first night after surgery. Acupuncture and moxibustion stimulation is applied to four pairs of acupoints: bilateral Shenmen (HT7), Neiguan (PC6), Zusanli (ST36) and Zhaohai (KI6), which are selected according to the previous systematic review and the summary of clinical experience . The pillow used is a disposable, sterile, stainless steel needle with a length of 40mm and a diameter of 0.25mm. In the acupuncture group, the acupuncture and moxibustion successively acupunctured four points with a depth of 10-20mm. Select the specific depth based on the subject's body type (tall, short, fat, thin). After the puncture, the acupuncture and moxibustion lifted and twisted the needle handle, and then retained the needle for 20 minutes. The sham acupuncture group received non skin breaking comfort needles at corresponding points for acupuncture and moxibustion the night before the operation, the night of the operation and the first night after the operation, and kept the needles for 20 minutes. Non transdermal comfort needles can cause patients to experience a needle like sensation similar to piercing the skin, but in reality, they do not break the skin. Before each application of acupuncture, it is necessary to evaluate whether the patient can perform acupuncture and moxibustion and whether there is a history of fainting. If there is a history of needle dizziness, the trial must be withdrawn.

ii. On the day before surgery, the first day after surgery, the second day, and the day before discharge, the sleep status should be continuously monitored using a sleep monitoring screening device (ZG-S01D).

iii. The degree of postoperative acute pain mainly includes the pain during rest, activity, and coughing on the first to seventh day after surgery or during hospitalization (when hospitalization days are less than 7 days). The evaluation time point is twice a day (9am and 3pm) on postoperative days 1-2; From the 3rd to the 7th day after surgery, once a day (9am). Pain description and the impact of pain on body function should be evaluated once on the 7th day after surgery or discharge day. In addition, on the first day after surgery at 9am, patients were also asked to recall the most severe resting pain level after surgery; The degree of pain within 24 hours after surgery (1 hour, 4 hours, 8 hours, and 16 hours) is indirectly reflected by heart rate, blood pressure, and blood oxygen saturation (medical record review). The severity of postoperative acute pain in patients is mainly obtained by researchers through face-to-face pain assessment, with the assistance of nurses if necessary.

iiii. Postoperative chronic pain (CPSP) of patients and pain during follow-up include four aspects: pain incidence, pain description, pain severity, and the impact of pain on body function. The evaluation is mainly conducted by researchers through telephone follow-up, with evaluation times of 2 weeks, 1 month, 2 months, 3 months, and 6 months after surgery, respectively. The pain followed up at 3 months after surgery is postoperative chronic pain.

If you agree to participate in this study, please sign this informed consent form. During the entire study period, it is planned to collect 5 additional blood samples, each containing 5ml, with a total volume of approximately 25ml, for the determination of serum levels of IL-1, IL-6, TNF - α, plasma levels of 5-HT, DA, NE, and melatonin.

ELIGIBILITY:
Inclusion Criteria:

- Case selection: Patients undergoing elective thoracoscopic assisted radical resection for lung cancer, ASA grade I-II, aged 18-75 years.

Inclusion criteria:

1. Hospitalized patients aged ≥ 18 years old;
2. The surgical method is non emergency thoracoscopic assisted radical resection of lung cancer;
3. Patients with normal mental state, able to understand NRS scores, and correctly assess the degree of pain;
4. Patients who are informed and agree to the research objectives as explained.
5. Body Mass Index (BMI) 18.5-28 kg/m2
6. Preoperative clinical tumor lymph node metastasis (TNM) staging: according to cTis-3N01M0 of AJCC/UICC 8th edition.

Exclusion Criteria:

1. Patients with critical preoperative conditions or inability to cooperate;
2. Patients with postoperative disease recurrence, chronic infection, reoperation, or death;
3. Patients with severe complications, critical illness, or inability to cooperate after surgery;
4. Pittsburgh Sleep Quality Index (PSQI) score ≥ 7 or Insomnia Diagnosis - Ashens Insomnia Scale (AIS) score ≥ 6;
5. Sleep apnea or moderate or severe snoring;
6. In situ pacemaker, preoperative sinus bradycardia (heart rate ≤ 50 beats/minute) or sinoatrial node disease, second or third degree atrioventricular block
7. Long term use of anticonvulsants, antidepressants, or other psychotropic drugs
8. Severely sensitive or allergic to the drugs or devices in this study
9. Severe heart, liver, or kidney disease;
10. Participated in other clinical trials within the past 3 months;

h) Listening and/or language communication barriers; i) Pregnancy or breastfeeding; j) Clinical (hematological, radiological, and/or microbiological) evidence of fever (body temperature 38.5 ℃) or preoperative infection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 316 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of Postoperative Sleep Disorders as Assessed by sleep monitoring screening device (ZG-S01D) and The The Athens Insomnia Scale | From enrollment to the end of treatment at 1 week;
  The Athens Insomnia Scale (AIS) is a self-assessment scale designed based on the ICD-10 diagnostic criteria for insomnia. There are a total of 8 questions, with the first 5 questions evaluating nighttime sleep and the last 3 questions evaluating daytime function. The scoring range for each question is 0-3, with a total score of 24 points. A score greater than or equal to 6 indicates the presence of sleep disorders. AIS is suitable for evaluating sleep status in the past month.

CONTACTS AND LOCATIONS:
Overall Officials: Shanghai 1st, Study Director — Xueying Ding
Locations (1):
- Shanghai General Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No